CLINICAL TRIAL: NCT05742724
Title: The Pharmacokinetics of Oral Tetrahydrocannabinol and Cannabidiol Across the Spectrum of Glomerular Filtration Rate: a PharmacoKinetic Study
Brief Title: The Pharmacokinetics of Single Dose Oral Tetrahydrocannabinol and Cannabidiol
Acronym: POT-GFR-PK
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Center for Medicinal Cannabis Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: POT_GFR_PK_001
Record Dates: First submitted 2023-01-11; First posted 2023-02-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cannabis; Chronic Kidney Diseases; Dialysis
Keywords: Pharmacokinetics
MeSH Terms: conditions — Marijuana Abuse; Renal Insufficiency, Chronic | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THC/CBD (Experimental): Oral THC 0.1mg/kg and CBD 2.5mg/kg
  Interventions: Drug: Tetrahydrocannabinol-Cannabidiol Combination

INTERVENTIONS:
Drug: Tetrahydrocannabinol-Cannabidiol Combination — Oral THC 0.1mg/kg and CBD 2.5mg/kg

SUMMARY:
POT-GFR-PK is a single dose pharmacokinetic study oral tetrahydrocannabinol (THC) and cannabidiol (CBD) in healthy adult controls and individuals with chronic kidney disease including those treated with in-center hemodialysis.

DETAILED DESCRIPTION:
Adults aged greater than 25 years including 6 with eGFR>60ml/min/1.73m2, 6 eGFR 30-59ml/min/1.73m2, 6 eGFR <30ml/min/1.73m2 (CKD Epidemiology Collaboration equation) and 6 receiving in-center hemodialysis at least 2x weekly via a tunnelled catheter will receive THC 0.1mg/kg and CBD 2mg/kg by mouth in the form of MediPharm Labs-001 (MPL-001) (50mg CBD/2mg THC per 1mL). In healthy controls and participants with chronic kidney disease, blood samples will be collected at t=0, 1, 2, 3, 3.5 and 4 hours post THC/CBD administration. In participants receiving in-center hemodialysis, blood samples will be collected at t=0, 1, 2, 3, 3.5 and 4 hours post THC/CBD administration and during hemodialysis at t=0, 60, 120, 180 minutes and 15 minutes prior to the end of hemodialysis (at a reduced pump speed with blood flow 50-100ml/min) and 60 minutes post-hemodialysis. A 24 hour urine will be collected in all participants except those receiving hemodialysis without any residual urine output. Dialysate samples will be collected at 1,2,3 hours during hemodialysis and at the end of hemodialysis. Blood samples will also be collected at 24 and 48 hours. Plasma, urine and dialysis cannabinoids (THC, CBD and their metabolites) will be quantified using Multisegment Injection-Capillary Electrophoresis-Mass Spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. adult age>25 years
2. estimated glomerular filtration rate (eGFR)>60ml/min/1.73m2 or eGFR<60ml/min/1.73m2 by the CKD Epidemiology Collaboration equation including in-center hemodialysis at least 2x weekly for a minimum of 3 hours per treatment via a tunnelled catheter treated >90 days
3. agree to take the medication as directed in the study
4. provides informed consent

Exclusion Criteria:

1. body mass index <20 or >35kg/m2
2. physical dependence on any drug other than caffeine or nicotine
3. history of clinically significant adverse event associated with cannabis intoxication
4. history of psychosis or mania or any active major psychiatric disorder
5. recent (within 30 days) use of any cannabinoid (natural or synthetic) identified by self-report or urine drug screen for cannabinoids
6. taking any medication with known interactions with THC or CBD via cytochrome P450 (CYP) CYP2C9, CYP2C19 and CYP4A6 or CYP2D4 (e.g. anti-epileptic drugs, calcineurin inhibitors, anti-fungal)
7. evidence of liver dysfunction (ALT less than 3 times upper limit of normal, bilirubin below upper limit of normal, international normalized ratio<1.5)
8. pregnant or breastfeeding women
9. change in ideal body weight or dry weight in the last 4 weeks
10. intradialytic hypotension (systolic blood pressure<90mmHg) requiring an intervention in the previous 4 weeks

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Tetrahydrocannabinol and its metabolites maximum concentration (Cmax) | 48 hours
  Maximum concentration (Cmax)
Tetrahydrocannabinol and its metabolites time to Cmax | 48 hours
  Time to Cmax
Tetrahydrocannabinol and its metabolites last detection time | 48 hours
  Last detection time
Tetrahydrocannabinol and its metabolites area under the curve | 48 hours
  Area under the curve
Tetrahydrocannabinol and its metabolites renal clearance | 48 hours
  Renal clearance
Tetrahydrocannabinol and its metabolites dialytic clearance | 48 hours
  Dialytic clearance
Cannabidiol and its metabolites maximum concentration (Cmax) | 48 hours
  Maximum concentration (Cmax)
Cannabidiol and its metabolites time to Cmax | 48 hours
  Time to Cmax
Cannabidiol and its metabolites last detection time | 48 hours
  Last detection time
Cannabidiol and its metabolites area under the curve | 48 hours
  Area under the curve
Cannabidiol and its metabolites renal clearance | 48 hours
  Renal clearance
Cannabidiol and its metabolites dialytic clearance | 48 hours
  Dialytic clearance
Other cannabinoids and their metabolites maximum concentration (Cmax) | 48 hours
  Maximum concentration (Cmax)
Other cannabinoids and their metabolites time to Cmax | 48 hours
  Time to Cmax
Other cannabinoids and their metabolites last detection time | 48 hours
  Last detection time
Other cannabinoids and their metabolites area under the curve | 48 hours
  Area under the curve
Other cannabinoids and their metabolites renal clearance | 48 hours
  Renal clearance
Other cannabinoids and their metabolites dialytic clearance | 48 hours
  Dialytic clearance

SECONDARY OUTCOMES:
Adverse events | 48 hours
  Weakness, fatigue, pain, falls, abnormal coordination, numbness or tingling, sedation, sleepiness, tremor, confusion, disorientation, dissociation, abnormal speech, muscle spasms, nausea, vomiting, diarrhea, altered mood, depression, euphoric mood, hallucinations, blurred vision, dizziness, imbalance, palpitations, hypotension, syncope, urinary tract infection, allergic reactions, shortness of breath, lung infection, fever, sweatiness, headache
Blood pressure | 48 hours
  Systolic and diastolic blood pressure in mmHg
Heart rate | 48 hours
  Heart rate in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Michael Walsh, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No